CLINICAL TRIAL: NCT01849029
Title: Cognitive Processing Intervention for HIV/STI and Substance Use Among Native Women
Brief Title: Cognitive Processing Intervention for Trauma, HIV/STI Risks, and Substance Use Among Native Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cynthia Pearson, Research Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 43091-G; R34DA034529 (NIH)
Record Dates: First submitted 2013-05-04; First posted 2013-05-08 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Post Traumatic Stress Disorders; Unsafe Sex; Substance Use Disorders
Keywords: Post traumatic Stress Disorders; PTSD; HIV risk; sexual risk; substance use; alcohol misuse; Substance Abuse; Substance Addiction; Substance Dependence; Substance Use Disorders; Alcohol-Related Disorders; Binge Drinking; Sexual Partners; Sexual Behavior; Unsafe Sex
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Unsafe Sex; Substance-Related Disorders; Alcohol-Related Disorders; Binge Drinking; Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Processing Theapy-Cognitive (Experimental): Immediate group receives Cognitive Processing Therapy-Cognitive CPT-C intervention within one week of being consented into the study
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive
- Cognitive Processing Threapy-Cognitive (Other): Wait list group: waits 6 weeks before receiving the Cognitive Processing Therapy-Cognitive (CPT-C) intervention. During this period no intervention is received
  Interventions: Behavioral: Cognitive Processing Therapy-Cognitive

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy-Cognitive — Cognitive Processing Therapy-Cognitive (CPT-C) uses education about trauma reactions, emotional processing, and cognitive strategies to reduce trauma-related cognitive distortions. CPT is a manualised 12 session cognitive behavioral treatment for PTSD which offers an alternative to purely exposure based interventions. CPT has a smaller exposure component than imaginal exposure therapy and is therefore potentially more acceptable to clients or practitioners seeking alternatives to purely exposure focused treatments. CPT-C omits the written trauma account, and includes more practice of cognitive techniques during the sessions. The treatment was developed for twice weekly sessions over 6 weeks. It also directly targets associated problems such as depression, guilt and anger.
  Other Names: Cognitive Processing Therapy - Cognitive (CPT-C)

SUMMARY:
Many American Indian (AI) women never receive services for serious mental health problems resulting from traumatic events, violence exposure and maltreatment. AI women suffer higher lifetime rates of Post-traumatic Stress Disorder (PTSD) (20-23%), that often co-occur with excessive drinking and risky sexual behaviors. These factors magnify risk for human immunodeficiency virus and sexually transmitted disease (HIV/STI). In full development with tribal partners, this application, proposes a 3-year project to culturally adapt and pilot an empirically supported trauma-focused treatment, Cognitive Processing Therapy (CPT) for PTSD, substance use and HIV/STI sexual risk behavior among 50 AI women. Additionally, the investigators will assess the feasibility, acceptability and treatment fidelity of delivering CPT via AI community health workers in a resource-limited tribal reservation. This project brings a culturally responsive intervention to an understudied and highly vulnerable population. Its significance lies in its potential to advance science in the area of PTSD, substance use treatment and HIV/STI prevention among AI women. Study data would benefit tribal and rural communities and the mental health field. Finally, it is geared toward developing the research infrastructure and mental health treatment capacity serving AI women living in rural settings, a group at risk for an expanding HIV/AIDS epidemic. If successful, findings from this pilot will provide evidence for a larger effectiveness trial.

The AIMS are AIM I. Adapt the evidence-based CPT intervention in full collaboration with tribal partners. This will be done in accordance with the CDC's Map of Adaptation Process and involves formative research with tribal leaders, potential consumers, providers, and health care administrators using qualitative methodology.

AIM 2. Assess this intervention delivered by Native American community health workers for feasibility and acceptability in a resource-limited rural reservation setting.

AIM 3. Conduct a two-group, single-site waitlist randomized controlled pilot trial of a 12-session, 6-week CPT intervention among 56 (6 pilot) sexually active and substance using AI women with PTSD or sub-threshold PTSD. Determine preliminary efficacy and estimate an effect size in terms of three primary outcomes: (a) PTSD symptomatology; (b) substance use; (c) high risk sexual behavior.

DETAILED DESCRIPTION:
Nearly one of three American Indian (AI) women can expect to be raped in their lifetime putting them at great risk for revictimization and human immunodeficiency virus (HIV). The high prevalence of sexual and physical assault in Indian country has led Amnesty International to declare a state of emergency for AI women in the United States. This application is part of a community led effort by the Yakama Nation to turn this tide in their tribal community.

Situated in the plateau region of Eastern Washington, the Yakama Nation is the largest tribe in Washington State (comprising over 10,000 members.) Since 2008, Investigators at the University of Washington have been collaborating with the Yakama Reservation Wellness Coalition who has mobilized activists and researchers through a community-based participatory research (CBPR) process to address the trauma and associated mental health concerns disproportionately affecting community women. This application, in response to "R34 PA-09-146: Pilot and Feasibility Studies in Preparation for Drug Abuse Prevention Trials" proposes a 3-year project to culturally adapt and pilot an empirically supported trauma-focused treatment, Cognitive Processing Therapy (CPT) for post-traumatic stress disorder (PTSD), substance use and HIV/STI sexual risk behavior among 56 AI women in a resource-limited rural area.

Additionally, the investigators will assess the feasibility, acceptability and treatment fidelity of delivering this CPT via AI community health workers. Based on the investigators promising preliminary work, their multidisciplinary collaboration includes experienced AI and non-AI HIV, trauma, health service, and mental health academic researchers and an 8-member community research team of Yakama Nation tribal leaders, potential consumers, and health care providers with strong community connections.

High rates of comorbidity between substance and alcohol use disorders (SAUD) and PTSD have been well established especially for women. Moreover, 25-40% of those seeking treatment for substance use meet criteria for PTSD. Additionally, PTSD is associated with increased HIV-risk sexual behavior (HRSB) in women. Prevailing theory suggests that alcohol and other drugs may be used to self-medicate or mitigate PTSD symptoms, which then reinforces more substance use leading to substance abuse-related consequences and problems, particularly HIV/STI exposure. Avoidance of trauma-related cues and affect including avoidance through substance use is thought to maintain PTSD and enhance risky sexual behavior. Therefore, treatment of PTSD should decrease substance use and risky sexual behavior.

Many AI women never receive services for serious mental health problems resulting from traumatic events, violence exposure and maltreatment. AI women suffer higher lifetime rates of PTSD (20-23%), and are 2-3 times more likely than the general U.S. population to engage in excessive drinking which often co-occurs with risky sexual behaviors. These factors magnify risk for HIV and sexually transmitted infections (HIV/STI).

This project is innovative in both its focus and its methods. It brings a culturally responsive intervention to an understudied and highly vulnerable population. It will culturally adapt and modify an evidence-based community health worker delivered intervention to address health risk behaviors (SAUD and HRSB). Its significance lies in its potential to advance science in the area of PTSD and SAUD treatment and HIV/STI prevention among AI women. Study data would be a significant contribution to tribal and rural communities and the mental health field. Finally, it is geared toward developing the research infrastructure and mental health treatment capacity serving AI women living in rural settings, a group at risk for an expanding AIDS and STI epidemic. If successful, findings from this study will inform a larger efficacy trial.

AIM I. Adapt the evidence-based CPT intervention in full collaboration with tribal partners. This will be done in accordance with the CDC's Map of Adaptation Process and involved formative research with tribal leaders, potential consumers, providers, and health care administrators using qualitative methodology.

AIM 2. Assess this intervention delivered by Native American community health workers for feasibility and acceptability in a resource-limited rural reservation setting.

AIM 2. Conduct a two-group, single-site waitlist randomized controlled pilot trial of a 12-session, 6-week CPT intervention among 56 (6 pilot) sexually active and substance using AI women with PTSD or sub-threshold PTSD. Determine preliminary efficacy and estimate an effect size in terms of three primary outcomes: (a) PTSD symptomatology; (b) substance use; (c) high risk sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* Current Substance Use At least 2 days of heavy drinking in the past 30 day period (4 or more drinks over the course of 2 hours) OR Recent substance consumption (other than opioids) in the last 3 months
* Desire to abstain from substances
* Current Diagnostic and Statistical Manual -IV diagnosis of Post-traumatic stress disorder symptoms [score 30 or hire on the PTSD Checklist (PCL]
* Sexually active (past 12 months)
* Age ≥ 18 years
* Capacity to provide informed consent

Exclusion Criteria:

* Unstable psychiatric medication regimen (i.e., medication changes or dose changes in the past 2 months)
* Recent use of opioids (past 3 months)
* Current trauma-focused mental health treatment (MH) in the past 30 days
* Suicide attempt or suicidal ideation with intent or plan, or self-harm in the past month
* Presence of a psychotic disorder or uncontrolled Bipolar Disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Scale interview (PSS-I) | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  Post-traumatic stress disorder symptom severity scale range from 0 (no PTSD symptoms) to 51 (high PSTD symptoms); units on a scale
PTSD Symptom Scale interview (PSS-I) | Change from baseline (week 0) to follow-up (week 12-14)
  Post-traumatic stress disorder symptom severity scale range from 0 (no PTSD symptoms) to 51 (high PSTD symptoms); continuous, units on a scale

SECONDARY OUTCOMES:
Drug use Frequency (DUF) | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  DUF is a self-report measure of illicit drug use, rating what drugs were used, how often, and by which methods (injection, smoking, e.g.). Participant rates each drug on the same 0-7 frequency scale for the past 6 months (0=never, 1=several times, 2=about once a month, 3=several times a month, 4=1-2 days a week, 5=3-4 days a week, 6=5-6 days a week, 7=everyday)
Drug use Frequency (DUF) | Change from baseline (week 0) to follow-up (week 12-14)
  DUF is a self-report measure of illicit drug use, rating what drugs were used, how often, and by which methods (injection, smoking, e.g.). Participant rates each drug on the same 0-7 frequency scale for the past 6 months (0=never, 1=several times, 2=about once a month, 3=several times a month, 4=1-2 days a week, 5=3-4 days a week, 6=5-6 days a week, 7=everyday)
Short Inventory of Problems - Alcohol and Drugs, (SIP-AD) | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  SIP-AD 15-Item scale as a measure of consequence (0 no consequences to 45 high consequence)
Short Inventory of Problems - Alcohol and Drugs, (SIP-AD) | Change from baseline (week 0) to follow-up (week 12-14)
  SIP-AD 15-Item scale as a measure of consequence (0 no consequences to 45 high consequence)
Condom-protected sex | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  condom use is calculated by subtracting the number of vaginal or anal condom-protected sex acts in the last 6 weeks from the total number of sex acts then dividing the sum by the number of total sex acts.
  A continuous measure and dichotomous measure (at 100% condom use) will be assessed to report
Condom-protected sex | Change from baseline (week 0) to follow-up (week 12-14)
  condom use is calculated by subtracting the number of vaginal or anal condom-protected sex acts in the last 6 weeks from the total number of sex acts then dividing the sum by the number of total sex acts.
  A continuous measure and dichotomous measure (at 100% condom use) will be assessed to report

OTHER OUTCOMES:
Penn Alcohol Craving Scale (PACS) | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  a five-item self-administered instrument for assessing craving. Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking.
Penn Alcohol Craving Scale (PACS) | Change from baseline (week 0) to follow-up (week 12-14)
  a five-item self-administered instrument for assessing craving. Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking.
number of sex partners | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  count, dichotomized at one partner vs. more than one partner
number of sex partners | Change from baseline (week 0) to follow-up (week 12-14)
  count, dichotomized at one partner vs. more than one partner
sex under the influence of substances | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  1 item drank alcohol/ drug use before having vaginal or anal sex (yes/no)
sex under the influence of substances | Change from baseline (week 0) to follow-up (week 12-14)
  1 item drank alcohol/ drug use before having vaginal or anal sex (yes/no)
concurrent sexual partners | Change from baseline (week 0) to Post intervention (week 6-8 weeks)
  Overlapping partnerships where sexual (anal or vaginal) intercourse with one partner occurs between two acts of intercourse with another partner
concurrent sexual partners | Change from baseline (week 0) to follow-up (week 12-14)
  Overlapping partnerships where sexual (anal or vaginal) intercourse with one partner occurs between two acts of intercourse with another partner

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Pearson, PhD, Principal Investigator — Indigenous Wellness Research Institute, University of Washington
Locations (1):
- Yakama Nation Behavioral Health and Comprehensive Community Alcoholism Program and Youth Treatment Program, Toppenish, Washington, United States